CLINICAL TRIAL: NCT01455779
Title: Lyrette: Renewing Continence Objective and Subjective Efficacy Study
Acronym: ROSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Verathon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-3375
Record Dates: First submitted 2011-10-13; First posted 2011-10-20 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2013-11

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; Incontinence; SUI; Renessa
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lyrette (Other): The Verathon Transurethral RF System (Lyrette® System) is indicated for the treatment of female urinary stress incontinence (SUI) due to hypermobility in women who have failed conservative treatment and who are not candidates for surgical therapy.
  The treatment is a 9 minute non-surgical procedure completed using local anesthesia during a single office visit. Women are discharged home with no incisions, dressings, or catheters immediately following treatment.
  Interventions: Device: Lyrette

INTERVENTIONS:
Device: Lyrette — The Verathon Transurethral RF System (Lyrette® System) is indicated for the treatment of female urinary stress incontinence (SUI) due to hypermobility in women who have failed conservative treatment and who are not candidates for surgical therapy.
  The treatment is a 9 minute non-surgical procedure completed using local anesthesia during a single office visit. Women are discharged home with no incisions, dressings, or catheters immediately following treatment.

SUMMARY:
The purpose of this study is to demonstrate the treatment efficacy of the Lyrette® System in women most likely to be treated in an office setting for the condition of stress urinary incontinence, secondary to urethral hypermobility.

DETAILED DESCRIPTION:
This is a prospective, open-label, single arm clinical study to evaluate the Lyrette System (formerly Renessa System) in a population likely to be treated in a physician's office.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 60 years
* Female gender
* Ability to complete all study requirements
* Body Mass Index ≤ 35
* Incontinence Quality of Life score (IQOL) ≥ 55
* Leak Point Pressure (LPP) ≥ 90 cm H2O and
* Maximal Urethral Closure Pressure (MUCP) ≥ 45 cm H2O
* 3 to10 stress leaks recorded in the 3 day voiding diary
* Clinical history of stress urinary incontinence for ≥ 12 months
* Clinical diagnosis of stress urinary incontinence by study physician
* Clinical diagnosis of mixed incontinence with predominant stress component.
* Clinical diagnosis of bladder outlet hypermobility by a study physician
* Has failed conservative therapy (Kegels, biofeedback) and/or has not received conservative therapy for a period of at least 3 months prior to enrollment in the study.
* Medical Epidemiologic, and Social Aspects of Aging (MESA)stress symptom percentage score greater than urge symptom percentage score
* Post-void residual ≤ 100 cc with Stage II or lower pelvic organ prolapsed
* Urethral length ≥ 3 cm
* Is not a current smoker
* If subject has children, at least 1 year has elapsed after child birth and cessation of breastfeeding for at least 3 months, at enrollment.

Exclusion Criteria:

* ASA III or IV classification
* Current or planned pregnancy within the next 12 months
* Clinical diagnosis of detrusor overactivity by urodynamic evaluation
* Clinical diagnosis of mixed urinary incontinence with predominant urge component
* Clinical diagnosis of primary urge urinary incontinence
* Clinical diagnosis of gravitational loss
* Stage III, IV Pelvic Organ Prolapse
* Less than 2 grams of urine leakage during 1 hour stress pad test
* Previous surgery, RF micro-remodeling, or injection of bulking agents specifically for the treatment of urinary incontinence
* Current incontinence treatment with electrical stimulation, biofeedback, and/or medications
* Previous urethral and/or bladder surgery (excluding diagnostic endoscope)
* Current urinary tract infection
* History of chronic urinary tract infections
* History of recurrent pyelonephritis
* History of interstitial cystitis
* History of upper or lower urinary tract neoplasm
* History of upper or lower anatomic urinary tract abnormality or disorder
* History of acute or chronic renal failure
* Coagulopathy
* Immunosuppression (pathological or medication induced)
* Collagen vascular disease (scleroderma, etc.)
* Presence of a pacemaker, AICD, or other electrical health maintenance device, bladder neuro-modulation device.
* History of COPD or other obstructive pulmonary disease
* Life expectancy < 12 months
* Knowingly will be relocating out of practice area within 12 months of initiation of the study

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint will be assessed by the incidence of device related Serious Adverse Event's during the procedure and 30 days following treatment. | 30 days
  Safety will be assessed by the incidence of device related Serious Adverse Events's during the procedure and 30 days following treatment.
Primary Effectiveness Endpoint will be the proportion of "dry" patients at the 12 month follow-up. | 12 months
  The primary effectiveness endpoint will be the proportion of "dry" patients at the 12 month follow-up.

SECONDARY OUTCOMES:
Secondary Safety Endpoint will be the evaluation of Adverse Events through all follow-up visits | 36 months
  The secondary safety endpoints will be the evaluation of Adverse Events through all follow-up visits.
IQOL Score | 36 months from baseline
  An increase in overall IQOL score from baseline to 36 months.
Pad Weight | 12 months
  A 50% reduction in the amount of urine leaked during a 1-hour pad weight test
Cough Test Results | 12 months
  A negative cough test

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Tri Valley Urology Medical Group, Murrieta, California
  - Center for Bladder Control, Arlington Heights, Illinois
  - Women's Health Institute of Illinois, Oak Lawn, Illinois
  - Female Pelvic Medicine and Urogynecology, Grand Rapids, Michigan
  - Dial Research, Tennessee Women's Care, Nashville, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia